CLINICAL TRIAL: NCT00154518
Title: The Role of Matrix Metalloproteinases in Orthodontic Treatment
Brief Title: The Role of Matrix Metalloproteinases (MMPs) in Orthodontic Tooth Movement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 9261701411
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Tooth, Impacted; Molar, Third
Keywords: orthodontic tooth movement; matrix metalloproteinase; Orthodontics
MeSH Terms: conditions — Tooth, Impacted | interventions — Orthodontics

INTERVENTIONS:
Procedure: Orthodontic treatment

SUMMARY:
The purpose of this study is to test whether the two MMPs can be up-regulated during orthodontic treatment. Alveolar bone samples will be collected from partially impacted third molars after orthodontic uprighting for different periods of time in volunteers.

DETAILED DESCRIPTION:
Long treatment time is a major factor causing high fees for orthodontic treatment. Patients would have dental caries or periodontitis resulting from improper oral hygiene care during this long treatment period. How to speed up the tooth movement which determines the duration of orthodontic treatment, can help more people to obtain good occlusion and esthetics. Orthodontic force on a tooth induces bone resorption on the compression side and bone deposition on the tension side, thus the bone remodels and then the tooth moves. Therefore, bone resorption is the rate-limiting step of a lengthy orthodontic treatment.

Bone resorption is a complex process. The mineral component is dissolved by acid from osteoclasts. On the other hand, the organic components are digested with proteolytic enzymes secreted from osteoblasts and osteoclasts. We focus on our study on specific proteases which can digest extracellular matrix, called matrix metalloproteinases (MMPs). Osteoblast-derived MMPs play an important role during initiation of bone resorption. However, the mechanism of its regulation is not clear. The past studies applied stretching or tension on single layer of cultured cells to characterize cellular response to the mechanical stimulation. Now we simulate part of the bone resorption process by cultivating osteocyte-like cells in three-dimensional collagen gel under periodical compression.

In a preliminary study, we focus on transcriptional changes of MMPs upon compression in an osteosarcoma cell line MG-63. Initial data form microarray indicated specific increase of two MMPs expression after one day of compression. This increased expression was specific because the levels of house-keeping genes (ex. Beta-actin or GAPDH) and bone-specific markers were unaltered. Therefore, we proposed that increased MMP expression of osteoblasts under compression is the first step for bone remodeling switching from synthesis to degradation of osteoid. In order to test this hypothesis, the following specific aims will be achieved:

1. To test whether these two MMPs can be up-regulated during orthodontic treatment. Alveolar bone samples will be collected from partially impacted third molars after orthodontic uprighting for different periods of time in volunteers. In situ hybridization and immunohistochemistry analysis for MMPs will reveal their roles in this physiological process.
2. To optimize the regulation by changing the magnitude and frequency of the pressure, and characterize the time table for these changes.

ELIGIBILITY:
Inclusion Criteria:

* Two mandibular third molars containing at least one mesially angular impaction with crown exposed to oral cavity

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-01; Study Completion 2005-12

PRIMARY OUTCOMES:
Tissue staining with antibody

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chen Yao, DDS, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Dentistry, National Taiwan University Hospital, Taipei, Taiwan